CLINICAL TRIAL: NCT05565170
Title: Digitally Supported Lifestyle Programme to Promote Brain Health Among Older Adults - the LETHE Pilot Trial
Brief Title: Digitally Supported Lifestyle Programme to Promote Brain Health Among Older Adults
Acronym: LETHE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Medical University of Vienna (Other); Karolinska Institutet (Other); University Of Perugia (Other); FH Joanneum Gesellschaft mbH (Industry); Foundation for Research and Technology - Hellas (FORTH) (Unknown); Infotrend Innovations Co Ltd (Unknown); Innovation To Grow (Unknown); Kaasa solution GmbH (Unknown); Lisbon Council (Unknown); Maastricht University (Other); Combinostics Oy (Unknown); Alzheimer Europe (Other); Extra Red s.r.l. (Unknown); Stichting EGI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 101017405
Record Dates: First submitted 2022-09-26; First posted 2022-10-04 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Impairment; Cognitive Decline; Dementia
Keywords: Prevention; Risk reduction; Brain health; Lifestyle intervention; Digital intervention; eHealth; Telemedicine
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomised 1:1 to two parallel arms:
  * structured ICT-assisted multimodal lifestyle intervention (intervention group)
  * self-guided multimodal lifestyle intervention (control group)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be actively told to what group they have been assigned (intervention or control). Outcome assessors will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Structured ICT-assisted multimodal lifestyle intervention (Active Comparator): Participants assigned to this study arm follow an intensive structured, digitally supported multimodal lifestyle intervention programme (combination of individual and group-based in-person consultations/sessions and digital activities in the LETHE mobile phone App). Intervention duration is 2 years.
  Interventions: Behavioral: Structured ICT-assisted multimodal lifestyle intervention
- Self-guided multimodal lifestyle intervention (Sham Comparator): Participants assigned to this study arm receive regular health advice in connection with the study visits (and through a simplified version of the LETHE mobile phone App), and are recommended and encouraged to independently implement healthy lifestyle changes that are suitable and fit in with their daily routine. Intervention duration is 2 years.
  Interventions: Behavioral: Self-guided multimodal lifestyle intervention

INTERVENTIONS:
Behavioral: Structured ICT-assisted multimodal lifestyle intervention — The structured lifestyle intervention programme, partly tailored and personalised to individual needs, covers the following domains: physical activity, nutrition, cognitive activity, cardiovascular risk management, social interaction, sleep, and relaxation / stress management. The programme includes regular scheduled in-person sessions (group-based + individual) which are supported with independent digital activities in the LETHE App. The App has features such as e.g., a cognitive training programme, on-demand exercise videos, calendar to schedule activities, advice and educational material, group chat, and possibility to set and monitor goals and self-monitor risk factors such as e.g., blood pressure.
  Arms: Structured ICT-assisted multimodal lifestyle intervention
Behavioral: Self-guided multimodal lifestyle intervention — Participants are advised to build their own healthy lifestyle programme based on standard healthy lifestyle advice that they will receive at individual consultations with the study physician/nurse as part of the study visits and through the simplified version of the LETHE app. The control group app does not include any structured / scheduled activities or personalised content.
  Arms: Self-guided multimodal lifestyle intervention

SUMMARY:
Previous research has shown that a healthy lifestyle, including a balanced diet, physical and social activity, and management of vascular risk factors can support both cardiovascular and brain health. In a landmark Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER), a multimodal lifestyle programme had clear benefits on older adults' cognition, functioning, and quality of life. The LETHE study utilises novel technologies and digital tools to deliver an optimised and more personalised FINGER-type multimodal lifestyle intervention.

A total of 160 digitally skilled older adults (age 60-77) with risk factors for dementia but without substantial cognitive impairment will be recruited in Austria, Finland, Italy, and Sweden. Participants will be randomly assigned in a 1:1 ratio to the structured ICT-assisted multimodal lifestyle program (intervention group) or a self-guided lifestyle program (control group). Duration of the study and the intervention is 24 months. The multimodal lifestyle program covers the following domains: physical activity, nutrition, cognitive activity, vascular risk management, social interaction, sleep, and relaxation. The structured intervention program follows a hybrid model where regular in-person, individual and group-based intervention activities led by professionals are supported with activities in the LETHE mobile phone application. The self-guided (control) group receives relevant health advice and is recommended and encouraged to independently implement healthy lifestyle changes that are suitable and fit in with their daily routine. Control group will have access to a simplified version of the LETHE app without any structured, scheduled activities or personalized content.

The primary objective of the LETHE trial is to test the feasibility of a digitally supported multimodal lifestyle program (i.e., retention rate, adherence to intervention), and assess change in dementia risk based on validated risk scores (CAIDE, LIBRA). Other objectives include testing the intervention effects on lifestyle and risk factors, cognition, function, health-related quality of life, health literacy, physical functioning, and dementia-related biomarkers. To this aim, a range of personal, lifestyle, and health-related data will be collected both actively and passively with the help of digital devices. Attitudes towards digital tools and experiences of trial participation will also be explored.

DETAILED DESCRIPTION:
The LETHE pilot trial is a 24-month multicentre parallel-group randomised controlled trial conducted in Finland (Finnish Institute for Health and Welfare, THL), Austria (Medical University of Vienna, MUW), Sweden (Karolinska Institute, KI), and Italy (University of Perugia, UPG). LETHE is an academic-led trial (funded by EU Commission) where all four clinical centers are jointly and equally responsible for the planning and conduct of the trial.

The recruitment goal is 160 participants (40 per country). Participants will be recruited e.g., through public announcements or advertisements (newspaper, social media) and at the local study centres. Interested individuals will first be pre-screened to check the key inclusion criteria related to e.g., age, digital skills and readiness, and risk factor profile (CAIDE dementia risk score). Persons who appear to meet the inclusion criteria (and no reasons for exclusion have arisen) are then invited for the actual screening assessment visit (organised remotely or in-person) where the eligibility criteria are checked in detail (including cognition). Exclusion criteria are assessed by a physician (for those who meet the inclusion criteria). Eligible individuals are invited to the baseline visit at the study centre. After completing all baseline assessments, participants are randomised in 1:1 ratio to the intervention group (structured ICT-assisted multimodal lifestyle intervention) and control group (self-guided multimodal lifestyle intervention). Randomisation will be balanced across sites.

At the beginning of the study, all participants receive an Android smartphone (unless they have already a compatible phone which they prefer to use), first with a simplified version of the LETHE App installed where participants can complete a set of outcome assessment questionnaires (e.g., lifestyle-related). After randomisation, a visit is booked to hand out the Fitbit smartwatch (different versions for the intervention and control groups) and install the full study version of the App (also different for the different groups). The App and the smartwatch are used for both active and passive data collection throughout the trial, and to support the intervention delivery. The intervention group will be offered a structured and tailored multimodal lifestyle programme (based on the FINGER model) including regular in-person (face-to-face and remote) counselling and sessions led by professionals, as well as independent digital activities in the LETHE App. Sessions and activities are related to the following intervention components: physical activity, nutrition, cognitive activity, vascular risk management and monitoring, social interaction, sleep, and relaxation/stress management. Recommendations and plans are tailored. The LETHE App, which has been designed by the LETHE consortium for this project, has features such as e.g., a cognitive training program, on-demand exercise videos, calendar to schedule activities, advice and educational material, group chat, and possibility to set and monitor goals and self-monitor risk factors such as e.g., blood pressure. Participants in the self-guided group are instructed to build their own lifestyle programme based on general health and lifestyle recommendations that they will receive at the main study visits. They will also have access to a simplified version of the LETHE App with static educational content about healthy lifestyle, but without any structured and scheduled activities, interactive features, or personalised content.

After baseline, all participants are invited to the study centre for three main study visits to collect outcome information, at month 6, 12, and 24. The outcome assessors are blinded to the group allocation and participants are not actively told to which group they were assigned. Data collection through the digital devices takes place continuously. The primary objective of the trial is to assess the feasibility of the digitally supported multimodal lifestyle intervention programme, i.e., assess retention rate (what proportion of participants completes the 24-month intervention period) and adherence to the intervention and engagement with the digital tools. Furthermore, changes in validated dementia risk scores (CAIDE, LIBRA) are assessed. Other objectives include testing the intervention effects on lifestyle and different risk factors of cognitive decline and dementia, cognitive performance, physical functioning, health-related quality of life, health literacy, and dementia-related fluid and imaging biomarkers. Participants' experiences of study participation and views on e.g., the usability and acceptability of the digital tools will also be explored (through interviews/focus groups).

ELIGIBILITY:
Inclusion Criteria:

* Age 60-77 years
* Cardiovascular Risk Factors, Aging and Incidence of Dementia (CAIDE) Risk Score ≥ 6 points
* Cognitive performance at the mean level or slightly lower than expected for age, assessed with Mini-Mental State Examination (MMSE) and the Consortium to Establish a registry for Alzheimer's Disease (CERAD) verbal learning test (word list learning/recall)
* Proficiency in the local language (German, Italian, Finnish or Swedish)
* Ability and willingness to use an Android smartphone, access to and ability to use the internet (digital readiness)
* Existing compatible smartphone (Android) or willingness to use a new Android smartphone provided from the study

Exclusion Criteria:

* Dementia or substantial cognitive impairment (e.g., memory clinic referral needed as judged by the study physician)
* Current or past use of medications for Alzheimer's disease or related diseases (e.g., cholinesterase inhibitors, memantine)
* Diminished decision-making capacity, not capable of consenting or completing study assessments, based on clinical judgement
* Other significant neurologic disease, including but not limited to Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma with persistent neurologic sequelae or known structural brain abnormalities
* Any condition affecting safe engagement in the intervention, e.g., malignant disease, major depression, symptomatic cardiovascular disease, revascularisation within 1 year previously
* Severe loss of vision, hearing, or communicative ability; conditions preventing cooperation as judged by the study physician
* Concomitant participation in an interventional trial (unless this will not interfere with the LETHE trial based on study staff's judgement)

Ages: 60 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: retention rate | 24 months
  Percentage of participants completing the 24-month trial period in each study arm. Higher percentage indicates a better outcome.
Feasibility: adherence to the structured multimodal lifestyle intervention | Continuously measured during 24 months
  Attendance at scheduled intervention sessions (percentage), usage of / engagement with the digital devices (LETHE App, Fitbit smartwatch). Possible values range from a minimum of 0, with higher values indicating better adherence and more active engagement.
Change in dementia risk scores (LIBRA and CAIDE), units on a scale | Baseline, 12 months, 24 months
  Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) risk score and Change in the LIfestyle for BRAin health (LIBRA) score are validated tools to estimate late-life dementia risk based on a combination of non-modifiable and modifiable risk factors (CAIDE) or modifiable factors only (LIBRA). Total score ranges from 0 to 15 (CAIDE) and from -5.9 to +12.7 (LIBRA). Higher scores indicate higher risk.

SECONDARY OUTCOMES:
Change in healthy lifestyle, unit on a scale | Baseline, 12 months, 24 months
  Change in Healthy Lifestyle Index (brief score developed in the FINGER trial), a composite score based on self-reported data on exercise, diet, vascular factors, and cognitive/social activity (range 0-24, with a higher score indicating a better outcome)
Change in cognition: composite z-score based on an extended Neuropsychological Test Battery (NTB), unit on a scale | Baseline, 12 months, 24 months
  The NTB used in this study is adapted from the FINGER trial and includes the following tests:
  * Wechsler Memory Scale Revised, WMS-III, WMS-R, logical memory, immediate
  * WMS-R logical memory, delayed
  * WMS-R visual paired associates, immediate
  * WMS-R visual paired associates, delayed
  * WMS-R Digit Span, total
  * Rey Auditory Verbal Learning Test, RAVLT, learning (free recall)
  * RAVLT, delayed recall
  * CERAD category fluency
  * Category fluency (fruits and vegetables)
  * Trail Making Test (TMT) A
  * Trail Making Test (TMT) B, shifting score B-A
  * Stroop Test, shortened 40-stimulus version, condition 2
  * Stroop Test, condition 3, interference score 3 - 2
  * Wechsler Adult Intelligence Scale (WAIS) Digit Symbol Substitution Test (DSST)
  Higher z-score indicates better outcome (better cognitive performance).
Change in stress-related symptoms (Perceived Stress Scale, PSS-14), unit on a scale | Baseline, 12 months, 24 months
  PSS is a 14-item self-report scale assessing stress-related symptoms. Values ranging 0-56, with lower scores indicating a better outcome.
Change in sleep problems (Insomnia Severity Index, ISI), unit on a scale | Baseline, 12 months, 24 months
  The Insomnia Severity Index (ISI) is a validated seven item assessment tool to assist in the clinical evaluation of insomnia complaints. Values ranging 0-28, with lower scores indicating a better outcome.
Change in health-related quality of life (RAND-36), unit on a scale | Baseline, 12 months, 24 months
  The RAND-36 is comprised of 36 items that assess eight health concepts. The scale values are ranging 0-100, with higher scores indicating a better outcome.
Change in health literacy (short version of the European Health Literacy Survey Questionnaire, HLS-EU-Q16), unit on a scale. | Baseline, 24 months
  Health literacy will be assessed with the 16-item short version of the European Health Literacy Survey Questionnaire. Each item has four response categories (very difficult, fairly difficult, fairly easy and very easy), and higher scores indicate better health literacy.

OTHER OUTCOMES:
Exploratory: Change in physical activity - self-reported, unit on a scale | Baseline, 12 months, 24 months
  Self-reported physical exercise in the previous two weeks, using a modified version of the Minnesota Leisure Time Physical Activity Questionnaire, as number of sessions and average duration for each of the activities listed in the questionnaire. Higher levels of physical activity indicate a better outcome.
  Self-reported number of sessions of moderate-to-vigorous intensity exercise per week. A higher number of sessions indicates a better outcome.
Exploratory: Change in physical activity - objective, based on Fitbit smartwatch | Continuously for 24 months
  Objective measurement of physical activity levels, e.g., step count, using the Fitbit smartwatch which is worn continuously throughout the trial. Higher values indicate a better outcome.
Exploratory: Change in dietary intake, unit on a scale | Baseline, 12 months, 24 months
  A brief food frequency questionnaire is used to calculate scores reflecting adherence to a healthy diet (MEDAS score reflecting adherence to Mediterranean-type diet; Healthy Diet Index score developed in Finland in the context of FINGER and type 2 diabetes prevention studies). Higher scores indicate a better outcome.
Exploratory: Change in individual cognitive domains, unit on a scale | Baseline, 12 months, 24 months
  Composite z-scores for the:
  * memory
  * executive function
  * processing speed domains that are included in the NTB used as a measure for the primary outcome.
Exploratory: Change in cognition based on the digital assessment of cognitive performance (cCOG), unit on a scale | 1 month, 13 months, 25 months (approx. 1 month after each main study visit and NTB assessment)
  cCOG is a web-based self-administrable cognitive testing tool with three classical cognitive tasks: a modification of word list test, simple reaction task, and TMT. Higher scores and quicker performance indicate a better outcome.
Exploratory: Change in global cognition/function: Clinical Dementia Rating Sum of Boxes (CDR-SB), unit on a scale | Baseline, 24 months
  CDR and CDR Sum of Boxes (CDR-SB) scores are used to assess the influence of cognitive impairment on the ability to conduct everyday activities in patients with Alzheimer's disease and give a global clinical impression of the patient. CDR-SB Score values range from 0-18, with lower scores indicating better outcome.
Exploratory: Change in functioning level: Instrumental Activities of Daily Living (IADL), unit on a scale | Baseline, 12 months, 24 months
  Activity of Daily Living, Lawton-Brody Scale. Self-reported questionnaire assessing the level of functioning in eight daily activities necessary for living in the community. For each activity, the participant is rated either dependent (0 points) or independent (1 point). The score ranges 0-8, with a higher score indicating a better outcome.
Exploratory: Change in blood pressure, mmHg | Baseline, 6 months, 12 months, 24 months
  Changes in systolic and diastolic blood pressure, lower measurements indicate better outcomes
Exploratory: Change in Body Mass Index (BMI), kg/m² | Baseline, 6 months, 12 months, 24 months
  Calculated using baseline height, with lower BMI value indicating better outcome
Exploratory: Change in waist circumference, cm | Baseline, 6 months, 12 months, 24 months
  Lower waist circumference value indicating a better outcome
Exploratory: Change in concentration of blood lipids - total cholesterol, mmol/l | Baseline, 6 months, 12 months, 24 months
  Measured from serum, a lower total cholesterol value indicates a better outcome.
Exploratory: Change in concentration of blood lipids - HDL, mmol/l | Baseline, 6 months, 12 months, 24 months
  Measured from serum, a higher HDL value indicates a better outcome.
Exploratory: Change in concentration of blood lipids - LDL, mmol/l | Baseline, 6 months, 12 months, 24 months
  Measured from serum, a lower LDL value indicates a better outcome.
Exploratory: Change in concentration of blood triglycerides, mmol/l | Baseline, 6 months, 12 months, 24 months
  Measured from serum with lower triglycerides value indicating a better outcome.
Exploratory: Change in concentration of plasma glucose, mmol/l | Baseline, 6 months, 12 months, 24 months
  Measured from fasting blood sample, with lower glucose value indicating a better outcome.
Exploratory: Change in concentration of glycated haemoglobin (HbA1c), % | Baseline, 6 months, 12 months, 24 months
  Measured from fasting blood sample, with lower HbA1c value indicating a better outcome.
Exploratory: Change in heart rate, bpm | Continuously for 24 months
  Heart rate measured with Fitbit smartwatch
Exploratory: Change in amount of social interaction (based on the total count of nearby Bluetooth devices) | Continuously for 24 months
  Data on the total count of nearby Bluetooth devices collected via passive mobile phone sensors. Higher values indicate better outcome.
Exploratory: Change in physical functioning: timed 10-meter dual-task test, gait speed in m/s and gait cost | Baseline, 24 months
  Timed 10-meter dual task test combines a physical task (walking 10m) with a cognitive task (e.g., naming letters of the alphabet). The result is the time in seconds needed to complete this activity; gait speed is calculated in m/s. Shorter time and higher gait speed indicates a better outcome. Gait cost identifies the percentage of speed that is lost by adding a task to the walking and it is calculated as: GC= [(single-task gait velocity - dual-task gait velocity) / single-task gait velocity] × 100. Lower percentage indicates a better outcome.
Exploratory: Change in physical functioning: Short Physical Performance Battery (SPPB), unit on a scale | Baseline, 24 months
  Short Physical Performance Battery (SPPB) is a group of measures that combines the results of gait speed (score range 0-4), chair stand test (score range 0-4), and balance test (score range 0-4). The total score (sum of three domains) ranges from 0 to 12 (higher scores indicating better performance).
Exploratory: Change in physical functioning: hand grip strength, kg | Baseline, 24 months
  Hand grip strength using a handgrip dynamometer. Higher measures indicate a better outcome.
Exploratory: Change in depressive symptoms (Center for Epidemiologic Studies Depression Scale, CES-D), unit on a scale | Baseline, 12 months, 24 months
  The Center for Epidemiological Studies-Depression (CES-D) is a 20-item measure that asks how often over the past week symptoms associated with depression were experienced. Scores range from 0 to 60, with higher scores indicating greater depressive symptoms.
Exploratory: Change in sleep parameters based on Fitbit smartwatch data, unit on a scale | Continuously for 24 months
  Changes in quantitative and qualitative parameters of sleep (sleep stages, duration, and fragmentation) measured by the Fitbit smartwatch
Exploratory: Attitudes towards new technologies and novel digital solutions (System Usability Scale, SUS), unit on a scale | 1 month, 6 months, 24 months
  The SUS is a 10 item, widely used, psychometrically valid, and a simplified version is available for older adults with cognitive deficits. Scores are ranging 0-100 with higher scores indicating a better outcome.
Exploratory: Change in serum concentration of neurofilament light chain, NFL, pg/ml | Baseline, 24 months
  Blood levels of neurofilament light chain protein range from a minimum of 0, with lower levels indicating a better outcome.
Exploratory: Change in serum concentration of pTau-181, ng/uL | Baseline, 24 months
  Blood levels of phosphorylated tau-181 range from a minimum of 0, with lower levels indicating a better outcome.
Exploratory: Change in brain imaging markers: volumetry of brain segments based on magnetic resonance imaging, MRI | Baseline, 24 months
  Volumes of specific brain regions are assessed computationally.
Exploratory: Change in brain imaging markers: white matter lesions | Baseline, 24 months
  White matter lesion load is assessed computationally. Lower values indicate a better outcome.
Exploratory: Change in brain imaging markers: brain atrophy and vascular load, based on widely used rating scales, units on a scale | Baseline, 24 months
  Medial temporal lobe atrophy (MTA), global cortical atrophy (GCA) and Fazekas are assessed computationally. Lower scores indicate better outcomes.
Exploratory: Participant experiences of the trial and the usability, acceptability, and feasibility of the digital intervention tools | 24 months
  Qualitative data on the study experiences and opinions about the intervention and the LETHE App will be collected through interviews/focus groups with a subgroup of the intervention group participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tiia Ngandu, MD PhD, Principal Investigator — Finnish Institute for Health and Welfare; Elisabeth Stögmann, MD PhD, Principal Investigator — Medical University of Vienna; Francesca Mangialasche, MD PhD, Principal Investigator — Karolinska Institutet; Patrizia Mecocci, MD PhD, Principal Investigator — University Of Perugia
Locations (4):
- Medical University of Vienna, Vienna, Austria
- Finnish Institute for Health and Welfare, Helsinki, Finland
- University of Perugia, Perugia, Italy
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The LETHE consortium is open to requests from external researchers for data collected in this study. Applicants will be asked to submit a study protocol, including the research question, planned analysis, and data required. Data controllers will evaluate this plan (i.e., relevance of the research question, suitability of data, quality of proposed analyses, planned/ongoing LETHE analyses, and other matters) on a case-by-case basis and provide the data or reject the request. Shared data will encompass the data dictionary and de-identified data only. Any analysis will be conducted in collaboration with the LETHE Group. Access is subject to the LETHE legal framework. An access agreement will be prepared and signed by relevant parties.
Time Frame: Applications for data will be considered after the trial results have been published and data will be made available according to the terms of the access agreement.
Access Criteria: As described above in the Plan Description.

REFERENCES:
- [Derived] Rosenberg A, Untersteiner H, Guazzarini AG, Bodenler M, Bruinsma J, Buchgraber-Schnalzer B, Colombo M, Crutzen R, Diaz A, Fotiadis DI, Hilberger H, Huber S, Kaartinen N, Kassiotis T, Kivipelto M, Lehtisalo J, Loukas VS, Lotjonen J, Pirani M, Thunborg C, Hanke S, Mangialasche F, Mecocci P, Stogmann E, Ngandu T; on behaf of the LETHE Consortium. A digitally supported multimodal lifestyle program to promote brain health among older adults (the LETHE randomized controlled feasibility trial): study design, progress, and first results. Alzheimers Res Ther. 2024 Nov 21;16(1):252. doi: 10.1186/s13195-024-01615-4. PMID 39574193